CLINICAL TRIAL: NCT00390052
Title: A Phase I and Pharmacokinetic Study of Oral 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone(3-AP,Triapine) in the Treatment of Advanced Solid Tumors
Brief Title: 3-AP in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00139; NCI-2009-00139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-52; CDR0000507731; PHI-52 (Other: City of Hope); 7225 (Other: CTEP); U01CA062505 (NIH)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

ARMS (1):
- Arm I (Experimental): Patients will receive a 2-hour infusion of 3-AP once in week 1. Beginning in week 2, they will receive 3-AP by mouth twice a day 3 days a week for 3 weeks. Treatment with 3-AP by mouth may repeat every 4 weeks for as long as benefit is shown.
  Interventions: Drug: triapine; Other: pharmacological study; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: triapine — Given IV and orally
  Other Names: 3-AP; OCX-191
Other: pharmacological study — correlative study
  Other Names: pharmacological studies
Procedure: laboratory biomarker analysis — Correlative study

SUMMARY:
This phase I trial is studying the side effects and best dose of 3-AP in treating patients with advanced or metastatic solid tumors. 3-AP may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety, tolerability, and toxicity of oral 3-AP in patients with advanced solid tumors.

II. Determine the maximum tolerated dose and recommended phase II dose of this drug in these patients.

III. Determine the oral bioavailability and pharmacokinetics of this drug. IV. Assess tumoral expression of genes involved in response and resistance to 3-AP.

V. Observe and record any tumor response in these patients.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive a one time dose of 3-AP IV over 2 hours on day -7. Patients then receive oral 3-AP twice daily on days 1-3, 8-10, and 15-17. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of oral 3-AP until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Blood samples for pharmacokinetic analysis are collected periodically over 8 hours after the IV dose of 3-AP and after the first oral dose of 3-AP during course 1.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Criteria:

* Must be able to swallow
* Histologically confirmed solid tumor
* Advanced or metastatic disease
* Measurable or evaluable disease
* No known active CNS metastases
* ECOG performance status 0-1
* Life expectancy > 3 months
* Progressive disease during >= 1 prior standard therapy OR disease unlikely to respond to any currently available therapies
* Patients with previously treated CNS metastases who have no evidence of new CNS metastases AND are stable for >= 2 months are eligible
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL (transfusions allowed)
* Absolute neutrophil count >= 1,500/mm^3
* ALT and AST =< 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 times ULN
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 50 mL/min
* Bilirubin normal
* PT/PTT =< 1.5 times ULN
* FEV1 >= 1.2 L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 2 weeks prior to and during study treatment
* No mental deficits and/or psychiatric history that may preclude study treatment
* No active heart disease, including any of the following: myocardial infarction within the past 3 months, symptomatic coronary artery disease or heart block, uncontrolled congestive heart failure
* No moderate to severe compromise of pulmonary function
* No active infection
* No other life-threatening illness
* No active coagulation disorder other than occult blood
* No known positivity for glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Recovered from prior treatment
* Prior gemcitabine allowed
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 3 weeks since prior radiotherapy or any other treatment for this cancer
* No prior 3-AP
* No concurrent radiotherapy
* No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of oral 3-AP determined by dose-limiting toxicities graded according to the NCI CTCAE version 3.0 | 28 days

SECONDARY OUTCOMES:
Serum pharmacokinetics of oral triapine | Baseline, day 4, and day 8
  Summary statistics of the pharmacokinetic parameters will be tabulated using the logarithmic scale where appropriate. The relationship of the AUC to the dose will be assessed by least-square regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Yen, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States